CLINICAL TRIAL: NCT02367430
Title: Critical Time Intervention for Individuals With Hoarding Disorder
Acronym: CTI-HD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Carolyn I. Rodriguez, Associate Chair for Inclusion and Diversity in the Department of Psychiatry, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6681
Record Dates: First submitted 2015-02-13; First posted 2015-02-20 (Estimated); Results first posted 2020-02-11 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Hoarding Disorder
MeSH Terms: conditions — Hoarding Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Critical Time Intervention for Hoarding Disorder (Experimental): Patients with Hoarding Disorder received CTI Model
  Interventions: Behavioral: Critical Time Intervention With Buried in Treasures included

INTERVENTIONS:
Behavioral: Critical Time Intervention With Buried in Treasures included — Critical Time Intervention and BIT Workshop

SUMMARY:
The purpose of this study is to investigate whether a well-established case management model called Critical Time Intervention (CTI) can help individuals with hoarding disorder who are concerned about the risk of eviction. Each individual with hoarding disorder will be assigned to work with a CTI Specialist for 9 months, who will provide referrals for mental health treatment, legal consultations, and registration for entitlements. All participants will be offered a facilitated group intervention called the Buried in Treasures Workshop. The CTI Specialist will also facilitate reconnecting the individual with supportive family/friends and will monitor and support the de-cluttering of the patient's home.

ELIGIBILITY:
Inclusion Criteria:

* primary Hoarding Disorder
* age 18 or over
* Individuals concerned with the threat of eviction due to clutter
* Patient must be physically healthy
* Willing and able to understand and complete consent procedure
* English speaking

Exclusion Criteria:

* Not primary Hoarding Disorder
* Severly depressed patients; Hamilton depression rating scale greater than 30 or judged clinically to be at risk of suicide with Columbia Suicide Severity Rating Scale

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: H Blair Simpson, MD, PhD, Principal Investigator — Columbia-NYSPI-RFMH; Carolyn I Rodriguez, MD, PhD, Principal Investigator — Stanford University

REFERENCES:
- [Result] Millen AM, Levinson A, Linkovski O, Shuer L, Thaler T, Nick GA, Johns GK, Vargas SM, Rottier KA, Joyner E, Girson RB, Zwerling J, Sonnenfeld D, Shapiro AM, Tannen A, Conover S, Essock S, Herman D, Simpson HB, Rodriguez CI. Pilot Study Evaluating Critical Time Intervention for Individuals With Hoarding Disorder at Risk for Eviction. Psychiatr Serv. 2020 Apr 1;71(4):405-408. doi: 10.1176/appi.ps.201900447. Epub 2020 Jan 8. PMID 31910750

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study did not include a wash out or run in. Not applicable.
Period: Overall Study
Arm/Group | Critical Time Intervention for Hoarding Disorder
Started | 14
Completed | 11
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Critical Time Intervention for Hoarding Disorder
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Savings Inventory-Revised
Description: The Saving Inventory-Revised scale (SI-R) is a 23-item questionnaire with 3 factor-analytically defined sub-scales for difficulty discarding, excessive clutter, and compulsive acquisition.
  The total score (sum of 23 items) ranges from 0 to 92. Total score higher than 41 shows significant difficulty with clutter.
  For the acquisition subscale we sum items 2 (reverse score), 9, 11, 14, 16, 18 and 21. The subscale ranges from 0 to 28 and score greater than 13 indicates difficulty with excessive acquisition.
  For the difficulty discarding subscale we sum items 4(reverse score), 6, 7, 13, 17, 19, 23. The subscale ranges from 0 to 28 and score greater than 13 indicates difficulty with discarding.
  For the clutter subscale we sum items 1, 3, 5, 8, 10, 12, 15, 20, 22. The subscale ranges from 0 to 36 and score greater than 15 indicates difficulty with accumulated clutter.
Time Frame: Baseline, 3 months, 6 months and 9 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Critical Time Intervention for Hoarding Disorder
Number analyzed (Participants) | 14
units on a scale
  Baseline | 67.5 (2.5)
  3 months | 57.2 (4.1)
  6 months | 54.8 (5.2)
  9 months | 51.3 (4.6)

2. Primary Outcome: Clutter Image Rating Scale
Description: Clutter Image Rating ScaleL Three sets of photographs, each containing nine photos of a single room with varying levels of clutter. A selection is made as to which photograph best resembles their own home.
  This scale assesses the clutter levels in the bedroom, living room and kitchen. The scale for each room ranges from 1 to 9. Clutter that reaches the level 4 indicates significant difficulty with clutter that affects the person's life.
Time Frame: Baseline, 3 months, 6 months and 9 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Critical Time Intervention for Hoarding Disorder
Number analyzed (Participants) | 14
units on a scale
  Baseline | 6 (2)
  3 months | 5 (2)
  6 months | 5 (2)
  9 months | 5 (2)

ADVERSE EVENTS:
Time Frame: 9 months
Description: No adverse events were reported by participants
Arm/Group | Critical Time Intervention for Hoarding Disorder
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No